CLINICAL TRIAL: NCT01043900
Title: Right Prefrontal High Frequency rTMS in Treatment of Resistant OCD: a Double Blind, Randomized Controlled Trial
Brief Title: Efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) as an add-on Treatment for Resistant OCD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Carlos Gustavo Mansur, Department and Institute of Psychiatry, General Hospital, University of São Paulo Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: cgmansur01
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; rTMS; Transcranial Magnetic Stimulation; treatment; randomized controlled trials
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham rTMS (Placebo Comparator): Patients with stable medication regimen receiving 30 daily sessions of PLACEBO rTMS delivered to the right dorsolateral prefrontal cortex
  Interventions: Procedure: repetitive transcranial magnetic stimulation (rTMS)
- Active rTMS (Active Comparator): Patients with stable medication regimen receiving 30 daily sessions of active rTMS delivered to the right dorsolateral prefrontal cortex
  Interventions: Procedure: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Procedure: repetitive transcranial magnetic stimulation (rTMS) — 30 daily sessions: each with 40 trains of 5 seconds at 10Hz, with a 25 second inter-train interval, at an intensity of 110% of motor threshold. Site: Right Dorsolateral Prefrontal Cortex
  Other Names: TMS

SUMMARY:
OCD is a chronic condition with a high rate of poor responders to conventional treatments, such as antidepressants and psychotherapy. Chronic symptoms can lead to important social impairment and suffering for patients and families.

The present study aims to investigate if the addition of transcranial magnetic stimulation can provide enhanced response to conventional treatment.

Transcranial magnetic stimulation is a noninvasive technique that can influence specific areas of the brain and has very few side effects.

DETAILED DESCRIPTION:
The treatment with transcranial magnetic stimulation requires attendance to hospital daily sessions for 6 consecutive weeks. Each session lasts up to 30 minutes.

Side effects include scalp discomfort and mild headache. No anesthesia is required.

Stimulation aims the dorsolateral prefrontal cortex, a region previously studied to treat depression symptoms with positive results. The present technique has never been employed in previous studies, but risks are insignificant

ELIGIBILITY:
Inclusion Criteria:

* resistant OCD patients: maximum 25% reduction in Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) scores after at least 3 adequate trials with serotonin reuptake inhibitors (SRI) (including clomipramine) and 20 hours of cognitive behavioral therapy (CBT) or documented intolerance to either treatment.

Exclusion Criteria:

* metallic cerebral implants
* history of severe trauma or brain injury
* organic brain disease
* severe somatic disease
* history of drug dependence
* chronic psychosis
* present manic state

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
A reduction of at least 30 % in the Yale-Brown Obsessive Compulsive Scale (YBOCS) scores and an "improved" or "much improved" score on the Clinical Global Impression (CGI) improvement scale by the end of follow-up | 3 - 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos G Mansur, MD, Principal Investigator — Department and Institute of Psychiatry, General Hospital, University of São Paulo Medical School

REFERENCES:
- [Derived] Mansur CG, Myczkowki ML, de Barros Cabral S, Sartorelli Mdo C, Bellini BB, Dias AM, Bernik MA, Marcolin MA. Placebo effect after prefrontal magnetic stimulation in the treatment of resistant obsessive-compulsive disorder: a randomized controlled trial. Int J Neuropsychopharmacol. 2011 Nov;14(10):1389-97. doi: 10.1017/S1461145711000575. Epub 2011 Apr 18. PMID 21557884